CLINICAL TRIAL: NCT01733329
Title: Buccal Misoprostol During Cesarean Section for Preventing Postpartum Hemorrhage in Women With Risk Factors for Uterine Atony
Brief Title: Buccal Misoprostol During Cesarean Section for Preventing Postpartum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Flavio Hernández Castro, Principal Investigator, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GI07-011
Record Dates: First submitted 2012-11-16; First posted 2012-11-27 (Estimated); Results first posted 2014-03-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Postpartum Hemorrhage
Keywords: Buccal Misoprostol; Uterine Atony; Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia | interventions — Misoprostol; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to 400 mcg misoprostol (2 tablets) (n=60) placed in buccal space after umbilical cord clamping by anesthesiologist. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Interventions: Drug: Misoprostol
- Folic Acid (Placebo Comparator): women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to 10 mg Folic acid (2 tablets) (n=60) placed in buccal space after umbilical cord clamping by anesthesiologist. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Misoprostol — At cord clamping 2 tablets (400 mcg) were placed in the patient´s buccal space by anesthesiologist.
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Folic Acid — At cord clamping 2 tablets (10 mg) were placed in the patient´s buccal space by anesthesiologist.
  Other Names: Placebo
  Arms: Folic Acid

SUMMARY:
Objective: to demonstrate that buccal misoprostol administration during cesarean delivery in women with risk factors for uterine atony decreases the need for additional uterotonic medications, uterine atony and postpartum hemorrhage.

Design: randomized, double-blinded, placebo-controlled trial.

DETAILED DESCRIPTION:
Patients and methods: 120 pregnant women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to either 400 mcg misoprostol (n=60) or placebo (n=60) placed in buccal space after umbilical cord clamping. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent delivery either by elective or emergent cesarean section at 24 week gestation or later with preoperative levels of hemoglobin and hematocrit determined up to 72 hours prior to delivery. The patients must have at least one of the risk factors for uterine atony listed below:

  1. Fetal macrosomia (estimated fetal weight ≥ 4 Kilos) diagnosed by clinical measurement (Johnson´s technique) or ultrasound measurement (Hadlock´s formula).
  2. Polyhydramnios (defined as Phelan´s amniotic fluid index > 24 cm)
  3. Twin or Multiple pregnancy.
  4. Prolonged labour (prolonged active phase > 12 hours) or precipitate labour(cervical dilatation ≥ 10 cm/hour).
  5. Magnesium sulphate or any other tocolytic agent therapy for ≥ 8 hours before cesarean section.
  6. Intravenous oxytocin therapy for at least 4 hours before cesarean section.
  7. Multiparous women (≥ 3 prior abdominal or vaginal deliveries )
  8. Clinical chorioamnionitis was defined as maternal temperature of ≥ 38°C in addition to more than one of the following criteria: fetal tachycardia (> 160 beats per minute), maternal tachycardia (>100 beats per minute, maternal leukocytosis (15,000 cells/mm3), uterine tenderness or foul smelling amniotic fluid.
  9. Known myomatosis, uterine Müllerian malformations or those diagnosed by ultrasound.

Exclusion Criteria:

1. Misoprostol incorrect administration
2. Severe allergic, bleeding disorders (e.g., haemophilia); severe asthma or any other absolute contraindication to misoprostol use.
3. Any bleeding occurred before delivery (abruptio placentae, placenta praevia) or bleeding due to other causes different than uterine atony.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. José Eleuterio González, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Hamm J, Russell Z, Botha T, Carlan SJ, Richichi K. Buccal misoprostol to prevent hemorrhage at cesarean delivery: a randomized study. Am J Obstet Gynecol. 2005 May;192(5):1404-6. doi: 10.1016/j.ajog.2004.12.033. PMID 15902121
- [Derived] Hernandez-Castro F, Lopez-Serna N, Trevino-Salinas EM, Soria-Lopez JA, Sordia-Hernandez LH, Cardenas-Estrada E. Randomized double-blind placebo-controlled trial of buccal misoprostol to reduce the need for additional uterotonic drugs during cesarean delivery. Int J Gynaecol Obstet. 2016 Feb;132(2):184-7. doi: 10.1016/j.ijgo.2015.06.060. Epub 2015 Oct 23. PMID 26534874

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol: women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to either 400 mcg misoprostol (n=62) or placebo (n=61) placed in buccal space after umbilical cord clamping. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Misoprostol
- Folic Acid: women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to either misoprostol (n=60) or 10 mg Folic acid (n=60) placed in buccal space after umbilical cord clamping. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Placebo
Period: Overall Study
Arm/Group | Misoprostol | Folic Acid
Started | 62 | 61
Completed | 60 | 60
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Uterine artery injury | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Misoprostol: women with risk factors for uterine atony who underwent cesarean delivery assigned randomly to 400 mcg misoprostol (2 tablets) (n=60) placed in buccal space after umbilical cord clamping by anesthesiologist. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Misoprostol
- Folic Acid: women with risk factors for uterine atony who underwent cesarean delivery assigned randomly to 10 mg Folic acid (2 tablets) (n=60) placed in buccal space after umbilical cord clamping by anesthesiologist . The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Placebo
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Folic Acid | Total
Number analyzed (Participants) | 62 | 61 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.05 (5.32) | 25.18 (6.29) | 24.62 (5.83)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 4 | 11
  Between 18 and 65 years | 55 | 57 | 112
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 61 | 123
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 62 | 61 | 123

OUTCOME MEASURES:

1. Primary Outcome: Need for Additional Uterotonic Medications
Description: The surgeon requested additional uterotonic agents on the basis of the clinical findings during surgery (e.g. uterine atony or blood loss of at least 1000 mL) Additional oxytocin was considered additional oxytocic intervention for purposes of data analysis.
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Groups:
- Misoprostol: women with risk factors for uterine atony who underwent cesarean delivery were assigned randomly to either 400 mcg misoprostol (n=60) or placebo (n=60) placed in buccal space after umbilical cord clamping. The primary outcome variables were the need for additional uterotonic agents, estimated blood loss and uterine atony.
  Misoprostol
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 60 | 60
percentage of participants | 10 | 40
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p < 0.01, Fisher Exact

2. Secondary Outcome: Uterine Atony
Description: Uterine atony is defined as failure of the uterus to contract adequately following delivery. Recognition of a soft, "boggy" uterus in the setting of excessive postpartum bleeding can alert the attendant to atony and should trigger a series of interventions aimed at achieving tonic sustained uterine contraction.
Time Frame: 24 hours
Measure: Number; unit: percentage of participants
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 60 | 60
percentage of participants | 8.3 | 25
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p = 0.026, Fisher Exact

3. Secondary Outcome: Postpartum Hemorrhage
Description: Defined as:
  Estimated blood loss ≥1000 mL after cesarean delivery. A substantial fall in the haematocrit e.g. 10% The requirement for a blood transfusion
Time Frame: 24 HOURS
Measure: Number; unit: percentage of patients
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 60 | 60
percentage of patients | 6.6 | 20
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p = 0.058, Fisher Exact

4. Secondary Outcome: Blood Loss
Time Frame: 24 hours
Measure: Median (Standard Deviation); unit: mL
Arm/Group | Misoprostol | Folic Acid
Number analyzed (Participants) | 60 | 60
mL | 470 (149.91) | 653.33 (342.21)
Statistical Analysis 1: Comparison: Misoprostol vs Folic Acid; Test type: Superiority or Other; p = 0.007, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Misoprostol | Folic Acid
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
1. Technical problems with blood loss measurement leading to blood transfusion before receiving hematocrit result.
2. Small number of patients fulfill inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No